CLINICAL TRIAL: NCT04831398
Title: The Effects of Acute Melatonin Supplementation on Cardiovascular Responses to Sympathetic Activation
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Oklahoma (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 13084
Record Dates: First submitted 2021-04-01; First posted 2021-04-05 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Healthy
MeSH Terms: interventions — Melatonin

STUDY DESIGN:
Intervention Model Description: This study is a single-blind crossover design.
Who Masked: Participant
Masking Description: Participants will be blinded in two trials. Practitioners and operators will not be allowed to communicate with the participants concerning whether they are receiving placebo/melatonin. Outcome assessors and statisticians may not be blinded to experimental allocation. Our placebo should satisfy two conditions of an ideal placebo: a) it should be indistinguishable from the experimental supplement to blinded participants, and b) it should be physiologically inert. In this study, 1 microliter McCormicks Pure Mint Extract will be mixed with 29 ml of filtered water and given to participants as a sublingual spray. This mixture will be non-caloric and will mimic the taste and sensation of the commercially available melatonin spray that will be used in the study (Onnit Labs Inc., Mint Flavor).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo (PLA) is 10 sublingual sprays of a diluted (1 microliter/29ml filtered water) mint extract.
  Interventions: Other: Placebo
- Melatonin (Experimental): 5mg commercially available melatonin (MEL) spray will be given sublingually.
  Interventions: Dietary Supplement: melatonin

INTERVENTIONS:
Dietary Supplement: melatonin — A 5mg dose of melatonin spay will be delivered sublingually.
  Arms: Melatonin
Other: Placebo — 10 sprays of diluted mint extract. This mimics the sensation and taste of the melatonin spray
  Arms: Placebo

SUMMARY:
the purpose of this experiment is to determine if acute melatonin supplementation alters central and peripheral cardiovascular responses to a cold pressor test at rest and during dynamic exercise.

DETAILED DESCRIPTION:
After IRB approval, experiments will take place in the Human Circulation Research Laboratory in the Department of Health and Exercise on the University of Oklahoma Norman campus. All subjects will complete a total of 3 visits. The first is a screening visit to provide informed consent and to ensure the potential participant meets all inclusion criteria and no exclusion criteria. Once consented and enrolled, participants will be familiarized with experimental protocols. On separate days (visits 2 and 3), participants will complete placebo (PLA) and melatonin (MEL) in a randomly ordered, single-blind, counter-balanced design. PLA or MEL treatment will precede testing by 30min to maximize absorption into the circulation (Bartoli, 2013).

All experiments (PLA/MEL) will begin with the subject lying supine for 5 min of quiet rest where baseline measurements are taken, followed by activation of the lower body negative pressure (LBNP) device causing suction at -20 mmHg. Following LBNP participants will be given 10 minutes of rest to recover all variables to pre-LBNP values. After which participants will be given a hand grip dynamometer to complete 7 minutes of exercise at an intensity of 20% MVC at a 1s contraction to 2s relaxation cycle paced by a metronome. During the final 2 minutes of the 7 minutes of exercise the LBNP device will be activated again to -20mmHg such that the participant will be completing LBNP during rhythmic grip exercise. After the completion of exercise, the subject will remain supine for 10min. Then the a Total Labile Signal (TLS) procedure will be conducted. Where the experimental limb is occluded using a blood pressure cuff for 5min. The cuff is then rapidly deflated. The lowest oxyhemoglobin measured during the occlusion is recorded. After the TLS procedure, the subject will be de-instrumented and will leave the laboratory.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men and women
* Women must be premenopausal with a regular menstrual cycle (26-30 days)

Exclusion Criteria:

* History of autonomic dysfunction
* Cardiovascular diseases
* Diabetes
* Tobacco/nicotine use
* Systolic Pressure >= 130 mmHg
* Diastolic Pressure >= 85 mmHg
* Regular melatonin use >= 1 use/week
* Allergy to melatonin
* Cardiometabolic medication use (e.g. anti-hypertensives, insulin-sensitizing, statins)
* Sex hormone replacement medical use (e.g. testosterone, estrogen, progesterone)
* Pregnancy

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Muscle Tissue Oxygenation | 7 minutes of rest and 7 minutes of exercise
  Concentrations of Total, Oxy, and deoxyhemoglobin of Flexor Digitorum Profundus muscle of the forearm
Mean Arterial Pressure | 7 minutes of rest and 7 minutes of exercise
  average pressure within the arteries

SECONDARY OUTCOMES:
Cerebral Oxygenation | 7 minutes of rest and 7 minutes of exercise
  Concentrations of Total, Oxy, and deoxyhemoglobin of the Prefrontal Cortex of the brain
Heart Rate | 7 minutes of rest and 7 minutes of exercise
  number of heart beats per minute
Respiratory Rate | 7 minutes of rest and 7 minutes of exercise
  number of breaths per minute
Cardiac Output | 7 minutes of rest and 7 minutes of exercise
  volume of blood pumped by the heart per minute
Stroke Volume | 7 minutes of rest and 7 minutes of exercise
  volume of blood pumped by the heart per heart beat
Total peripheral resistance | 7 minutes of rest and 7 minutes of exercise
  amount of force affecting resistance to blood flow throughout the circulatory system
Heart Rate Variability | 7 minutes of rest and 7 minutes of exercise
  measure of the variation in time between each heart beat

CONTACTS AND LOCATIONS:
Overall Officials: Jeremy M Kellawan, Principal Investigator — University of Oklahoma
Locations (1):
- Department of Health and Exercise Science, Norman, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: No
The is no plan to share IPD